CLINICAL TRIAL: NCT00037596
Title: A Dose Ranging Study of the Safety and Efficacy of Gemtuzumab Ozogamicin (GO) Given in Combination With Cytarabine in Relapsed or Refractory Patients and Alder De Novo Patients With Acute Myeloid Leukemia.
Brief Title: Study Evaluating Gemtuzumab Ozogamicin in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 0903B1-205
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab; Cytarabine

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin
Drug: cytarabine.

SUMMARY:
The primary objectives are a) to establish the maximum tolerated dose of gemtuzumab ozogamicin in combination with cytarabine and b) to assess the safety of gemtuzumab ozogamicin when given concurrently with cytarabine.

ELIGIBILITY:
Inclusion Criteria:

* Morphologic diagnosis of AML from bone marrow aspirate and biopsy
* Flow cytometry, performed at the study site, must demonstrate that the patient has AML that is CD33+, based on local laboratory criteria
* Age 18 years or older for relapsed or refractory patients for Phase I of this study

Exclusion Criteria:

* Patients with de novo AML of the M3 subtype
* AML following an antecedent hematologic disorder (myelodysplasia or myeloproliferation) of > 2 months duration
* AML secondary to exposure to chemotherapy or radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Hibma J, Knight B. Population Pharmacokinetic Modeling of Gemtuzumab Ozogamicin in Adult Patients with Acute Myeloid Leukemia. Clin Pharmacokinet. 2019 Mar;58(3):335-347. doi: 10.1007/s40262-018-0699-5. PMID 30062662